CLINICAL TRIAL: NCT05514353
Title: A Phase 1, Randomized, Double-Blind, Vehicle-Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetic Characteristics of Single and Multiple Ascending Doses of PBI-100 Topical Cream in Healthy Adult Subjects and Subjects With Psoriasis
Brief Title: A Phase 1 Study to Assess Single and Multiple Ascending Doses of PBI-100 Topical Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PBI-100-102
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PBI-100 Topical Cream (Experimental): SAD: 4 cohorts of subjects are planned to receive a single dose of PBI-100 topical cream in one of three dosage strengths, administered once or twice daily
  MAD: 3 cohorts of subjects are planned to receive one of three dosage strengths of PBI-100 administered once or twice daily for periods of 14 consecutive days
  Interventions: Drug: PBI-100 Topical Cream
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: PBI-100 Topical Cream — PBI-100 Topical Cream in 1 of 3 dose levels
  Arms: PBI-100 Topical Cream
Drug: Vehicle Cream — The Vehicle Cream formulation contains the same excipients as the active cream
  Arms: Vehicle

SUMMARY:
This is a Phase 1, randomized, double-blind, vehicle-controlled, SAD / MAD study evaluating three dose levels of PBI-100 topical cream in healthy adult volunteers and/or subjects with psoriasis.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, vehicle-controlled, SAD / MAD study. Three dose levels of PBI-100 topical cream will be evaluated in healthy adult volunteers and/or subjects with psoriasis. Dose escalations will follow a satisfactory review by the Safety Review Committee of all available safety, tolerability, and PK data from the current dose level.

ELIGIBILITY:
Key Inclusion Criteria:

* Is male or female, between 18 and 65 years of age
* Has a body mass index (BMI) between 18.0 and 32.0 kg/m2
* Is in good general health, as determined by the Investigator, without clinically significant medical history, with the exception of psoriasis for those subjects enrolled in the psoriasis groups

Key Exclusion Criteria:

* Has any visible skin disease (other than psoriasis for subjects in Groups 4 and 7) at the application site which, in the opinion of the Investigator, would interfere with the evaluation of the test site reaction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) in Healthy Adult Subjects | From dosing until discharge, up to Day 28
  To assess safety and tolerability of single and multiple doses of PBI-100 Topical Cream
Number of Adverse Events (AEs) in Adult Subjects with Psoriasis | From dosing until discharge, up to Day 28
  To assess safety and tolerability of single and multiple doses of PBI-100 Topical Cream

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (1):
- TKL Research Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No